CLINICAL TRIAL: NCT01935323
Title: High Intensity Interval Versus Continuous Moderate Intensity Training: Maximizing the Benefits of Exercise in Overweight Adolescents.
Acronym: HIIT-MAX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: The Coca-Cola Company (Industry)
Responsible Party: Principal Investigator, David Allison, Phd, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: F121101004
Record Dates: First submitted 2013-06-20; First posted 2013-09-05 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 2016-01

CONDITIONS: Metabolism; Physical Fitness
Keywords: high intensity interval training; aerobic exercise; insulin sensitivity; obesity; cardiovascular fitness
MeSH Terms: conditions — Insulin Resistance; Obesity | interventions — High-Intensity Interval Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- High Intensity Interval Training (Experimental): Participants will perform the HIIT protocol on an electronically-braked cycle ergometer (Quinton Excalibur, Quinton Instrument Company, Bothell, WA). Participants will perform a 20-minute protocol, consisting of four minutes of cycling at 15% of maximum anaerobic power (Max-AP) followed by 30 seconds at 85% of Max-AP. These workloads will be based upon pre-trial Wingate tests. This cycle was repeated four times within each protocol, ending with two minutes at 15% of Max-AP. This will be performed 3d/wk for 6wks, with at least 24 hrs between each session.
  Interventions: Other: High Intensity Interval Training
- Moderate Intensity Training (Active Comparator): Participants will perform 45-60 min (graduated over time to 60) of continuous cycling at 65% of VO¬2peak on a Monark cycle ergometer. Workload will be based upon pre-trial VO¬2peak testing. MIT exercise will be performed 5d/wk for 6wks.
  Interventions: Other: Moderate Intensity Training

INTERVENTIONS:
Other: High Intensity Interval Training
  Arms: High Intensity Interval Training
Other: Moderate Intensity Training
  Arms: Moderate Intensity Training

SUMMARY:
6-week, single site, two parallel arm, randomized, controlled trial comparing the effectiveness of a High Intensity Interval Training (HIIT) versus a continuous Moderate Intensity Training (MIT) program on cardiovascular and metabolic health outcomes in overweight adolescent males. HIIT training may be a potent time-efficient strategy to induce similar metabolic and cardiovascular adaptations typically associated with MIT.

ELIGIBILITY:
Inclusion Criteria:

* Ages 17-22
* Men
* BMI (25.0 - 35.0 kg/m2)
* Interested in improving health and fitness

Exclusion Criteria:

* Weight loss or gain of >10% of body weight in the past 6 months for any reason.
* Currently taking medication that suppresses or stimulates appetite.
* History of prior surgical procedure for weight control or liposuction.
* Current smoker.

Any major disease, including:

* Active cancer or cancer requiring treatment in the past 2 years (except nonmelanoma skin cancer).
* Active or chronic infections, including self-reported HIV positivity and active tuberculosis.
* Diagnosed heart conditions.
* Uncontrolled hypertension: systolic blood pressure 160 mm Hg or diastolic blood pressure 95 mm Hg on treatment.
* Gastrointestinal disease, including self-reported chronic hepatitis or cirrhosis, any episode of alcoholic hepatitis or alcoholic pancreatitis within past year, inflammatory bowel disease requiring treatment in the past year, recent or significant abdominal surgery (e.g., gastrectomy).
* Asthma.
* Diagnosed diabetes (type 1 or 2), fasting impaired glucose tolerance (blood glucose 118 mg/dL), or use of any anti-diabetic medications.

  * Conditions or behaviors likely to effect the conduct of the trial: unable or unwilling to give informed consent; unable to communicate with the pertinent clinic staff; unwilling to accept treatment assignment by randomization; current or anticipated participation in another intervention research project that would interfere with the intervention offered in the trial; likely to move away from participating clinics before trial completed; unable to walk 0.25 mile in 10 minutes.
  * Currently taking antidepressant, steroid, or thyroid medication, unless dosage is stable (no change for 6 months).
  * Any active use of illegal or illicit drugs.
  * Excessive alcohol intake defined as an average consumption of 3 or more alcohol containing beverages daily.
  * Unwilling to limit alcohol intake to ≤2 drink per day (one drink = 4 oz. wine, 12 oz. beer, or ½ shot of liquor).
  * Current exerciser (>30 min organized exercise per week).
  * Indication of unsuitability of current health for exercise protocol (PARQ).
  * Any other conditions which, in opinion of the investigators, would adversely affect the conduct of the trial.

Ages: 17 Years to 22 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2013-02; Primary Completion 2014-10 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Body Composition as measured by DXA | Baseline and 6 weeks

SECONDARY OUTCOMES:
Body Weight | Baseline and 6 weeks
Blood Pressure | Baseline and 6 weeks
Body Mass Index | Baseline and 6 weeks
Peak uptake of volume of oxygen | Baseline and 6 weeks
Wingate Cycle test | Baseline and 6 weeks
LDL Cholesterol | Baseline and 6 weeks
HDL Cholesterol | Baseline and 6 weeks
Triglycerides | Baseline and 6 weeks
Glucose | Baseline and 6 weeks
Insulin | Baseline and 6 weeks
Ghrelin | Baseline and 6 weeks
Leptin | Baseline and 6 weeks
Adiponectin | Baseline and 6 weeks
PYY | Baseline and 6 weeks
IL-6 | Baseline and 6 weeks
TNF-alpha | Baseline and 6 weeks
Total antioxidant capacity | Baseline and 6 weeks
Protein Carbonyls | Baseline and 6 weeks
  ELISA assay purchased from NW LifeSciences. Prior to analysis, all serum samples were assayed for protein concentration based on the methods of Bradford and adjusted to 4 mg・mL-1 protein using a phosphate buffer. Protein carbonyls, a measure of protein oxidation, were analyzed in duplicate in 50 μl of sera using a commercially available ELISA kit (NWK-PCK01).The intra- and interassay coefficients of variation were 2.7 % and 5%. The lower detection limit of the assay was 0.1 nmol/mg.
Free living energy expenditure as measured by accelerometer | Baseline and 6 weeks
Appetite/satiety measures | baseline & 6 weeks
  composite score
Quality & satisfaction with life | baseline & 6 weeks
  composite score
Rate of perceived exertion during exercise via Borg Scale | baseline and 6 weeks
24-hour dietary recall | pre-baseline, baseline, 6 weeks
Self Motivation Inventory | baseline and 6 weeks
Profile of Mood States | baseline & 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- UAB Physiology Lab, Birmingham, Alabama, United States

REFERENCES:
- [Background] Fisher G, Brown AW, Bohan Brown MM, Alcorn A, Noles C, Winwood L, Resuehr H, George B, Jeansonne MM, Allison DB. High Intensity Interval- vs Moderate Intensity- Training for Improving Cardiometabolic Health in Overweight or Obese Males: A Randomized Controlled Trial. PLoS One. 2015 Oct 21;10(10):e0138853. doi: 10.1371/journal.pone.0138853. eCollection 2015. PMID 26489022
- See also: UAB Nutrition Obesity Research Center — http://www.norc.uab.edu